CLINICAL TRIAL: NCT05061017
Title: Phase IIA Basket Study of Pixatimod (PG545) in Combination With Nivolumab in PD-1 Relapsed/Refractory Metastatic Melanoma and NSCLC and Pixatimod (PG545) in Combination With Nivolumab and Low-dose Cyclophosphamide in MSS Metastatic Colorectal Carcinoma (mCRC)
Brief Title: Pixatimod (PG545) Plus Nivolumab in PD-1 Relapsed/Refractory Metastatic Melanoma and NSCLC and With Nivolumab and Low-dose Cyclophosphamide in MSS Metastatic Colorectal Carcinoma (mCRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Aculeus Therapeutics (Unknown)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-266
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: NSCLC; Metastatic Colorectal Carcinoma; Refractory Melanoma
Keywords: melanoma; PD-1/PD-L1 pathway; relapsed metastatic melanoma; refractory metastatic melonma; MSS Metastatic Colorectal Carcinoma; PD-1 R/R NSCLC; PD-1 R/R melanoma; MSS mCRC
MeSH Terms: conditions — Colorectal Neoplasms; Melanoma | interventions — PG 545; Nivolumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pixatimod (PG545) + Nivolumab (Experimental): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 (MSS CRC)
  Interventions: Drug: Pixatimod; Drug: Nivolumab
- Pixatimod (PG545) + Nivolumab + cyclophosphamide (Experimental): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Interventions: Drug: Pixatimod; Drug: Nivolumab; Drug: Cyclophosphamide (low dose)

INTERVENTIONS:
Drug: Pixatimod — Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Other Names: (PG545)
Drug: Nivolumab — Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Other Names: OPDIVO®
Drug: Cyclophosphamide (low dose) — Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
  Arms: Pixatimod (PG545) + Nivolumab + cyclophosphamide

SUMMARY:
The primary goal of this trial is to assess clinical response to nivolumab and pixatimod, and, nivolumab, pixatimod and cyclophosphamide in three separate patient cohorts. Cohort 1: MSS mCRC in combination with low-dose cyclophosphamide, Cohort 2: PD-1 relapsed/refractory melanoma, and Cohort 3: PD-1 relapsed/refractory NSCLC.

DETAILED DESCRIPTION:
Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer.

Pixatimod is an investigational drug that activates the toll-like receptor 9 (TLR9) pathway and is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.

Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab.

This Phase llA trial hypothesizes that the nivolumab/pixatimod combination in PD-1 relapsed/refractory (R/R) cutaneous melanoma and NSCLC patients will be associated with anti-tumor effects, and that the nivolumab/pixatimod/cyclophosphamide combination in MSS mCRC patients will be associated with anti-tumor effect.

In the 1st stage, 13 patients will be enrolled in cohort 1 while 9 patients each will be enrolled in cohorts 2 and 3. Should the pre-specified efficacy boundary met, further patients will be enrolled to one or more cohorts in 2nd stage. The total enrollment for 1st stage across all 3 cohorts is 31 response-evaluable patients. The total enrollment for both stages across all 3 cohorts is 61 response-evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Male/female participants who are at least 18 years of age on the day of signing informed consent with advanced/metastatic cutaneous melanoma, NSCLC or MSS mCRC who meet the following criteria will be enrolled in this study.
* Male participants:

  o A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants:

  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
  * Not a woman of childbearing potential (WOCBP);OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

Cohort 1 (MSS mCRC)

* MSS is defined as 0-1 allelic shifts among 3-5 tumor microsatellite loci using a PCR-based assay or immunohistochemistry.
* Must have received prior therapy with a fluoropyrimidine, oxaliplatin, and irinotecan.
* Prior treatment with an anti-PD-1/anti-PD-L1 or anti-CTLA-4 antibody is not allowed.
* Prior treatment with BRAF/MEK inhibitor therapy (if BRAF mutated) and/or EGFR targeted antibody (if KRAS WT) are allowed.
* No more than 2 prior lines of therapy for metastatic disease.
* Adjuvant therapy will count as 1 prior line of therapy if received within the prior 6 months; but if not does not count towards prior line of therapy.
* PIV (pan-immune-inflammation) cutoff of 1200 obtained on labs obtained during Screening.

Cohort 2 (PD-1 R/R melanoma)

* PD-1 refractory disease as defined as progression on treatment with anti-PD-(L)1 inhibitor administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

  * Receipt of at least 2 doses of an approved or investigational anti-PD-(L)1 inhibitor.
  * Demonstrated PD after anti-PD-(L)1 inhibitor as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression (as defined by the criteria in the sub-point below).
  * Progressive disease that has been documented within 12 weeks from the last dose of anti-PD-(L)1 inhibitor.
* Progressive disease is determined according to iRECIST.
* This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
* Subjects who progressed on/within 3 months of adjuvant therapy with anti-PD-(L)1 inhibitor will be allowed; an adjuvant therapy will count as 1 prior line of therapy if received within the prior 6 months.
* Prior treatment with an anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibody is allowed but not required.
* Prior treatment with BRAF/MEK inhibitor therapy (if BRAF mutated) is allowed but not required.
* No more than 5 prior lines of therapy.

Cohort 3 (PD-1 R/R NSCLC)

* PD-1 refractory disease as defined as progression on treatment with anti-PD-(L)1 inhibitor administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

  * Has received at least 2 doses of an approved or investigational anti-PD-(L)1 inhibitor.
  * Has demonstrated PD after anti-PD-(L)1 inhibitor as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression (as defined by the criteria in the sub-point below).
  * Progressive disease has been documented within 12 weeks from the last dose of anti-PD-(L)1 inhibitor.
* Progressive disease is determined according to iRECIST.
* This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
* Subjects who progressed on/within 3 months of adjuvant therapy with anti-PD-(L)1 inhibitor will be allowed; an adjuvant therapy will count as 1 prior line of therapy if received within the prior 6 months.
* Prior treatment with an anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibody is allowed but not required.
* Prior treatment with BRAF/MEK inhibitor therapy (if BRAF mutated) must have received and progressed or have demonstrable intolerance to approved targeted therapy.
* Patients with NSCLC with known oncogenic driver (including but not limited to EGFR, ALK, ROS, MET alterations) must have received and progressed past driver-specific therapy.
* No more than 5 prior lines of therapy.

Other Criteria

* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided newly obtained core or excisional biopsy of a tumor lesion not previously irradiated to undergo tumor biopsy (core, punch, incisional or excisional).

  o Biopsy must meet minimal sampling criteria.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 28 days prior to the date of enrollment.
* Adequate organ function. Screening labs obtained within 4 weeks of Cycle 1 day 1
* Proteinuria exceeding 1gram in a 24 hour period.
* A pan-immune-inflammation (PIV) cutoff of 1200 (obtained on labs during Screening)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* History of allergy and/or hypersensitivity and/or other clinically significant adverse drug reaction to heparin or other anti-coagulant agents, or to any monoclonal antibody.
* Use of heparin (including low-molecular weight heparin and/or fondaparinux) within 2 weeks prior to enrollment.

  o Patients who are currently receiving low-molecular weight heparin (or fondaparinux or other heparin product) for therapeutic anticoagulation may be enrolled if they have tested negative for anti-heparin antibodies at Screening.
* Has a diagnosis of immunodeficiency, immunosuppression and/or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  * Note: Subjects with autoimmune disorders of Grade 4 while on prior immunotherapy will be excluded. Subjects who developed autoimmune disorders of Grade ≤ 3 may enroll if the disorder has resolved to Grade ≤1 and the subject has been off systemic steroids at doses >10 mg/d for at least 2 weeks.
* Active (i.e., symptomatic or growing) central nervous system (CNS) metastases.

  * Note: Subjects with treated and stable CNS metastases are permitted to enroll. Stability for prior treated CNS disease should be assessed on a contrast-enhanced imaging study obtained no sooner than 14 days from data of definitive radiotherapy and/or surgery for CNS disease.
  * Note: Subjects with leptomeningeal carcinomatosis are excluded.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone (or is being planned to undergo) potentially curative therapy.
* Has a systemic disease that requires systemic pharmacologic doses of corticosteroids greater than 10 mg daily prednisone (or equivalent).

  * Note: Subjects who are currently receiving steroids at a dose of ≤10 mg daily do not need to discontinue steroids prior to enrollment.
  * Note: Subjects that require topical, ophthalmologic and inhalational steroids are not excluded from the study.
  * Note: Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome are not excluded from the study.
  * Note: Subjects who require active immunosuppression (greater than steroid dose discussed above) for any reason are excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 26 weeks after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

  o Note: Subjects with HIV that is well controlled (undetectable viral load and CD4 count >200 cells/mm3) on anti-retroviral therapy are permitted to enroll.
* Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected.

  o Note: Subjects with treated hepatitis B and/or C with no evidence of active infection may be enrolled.
* Has a history of significant cardiac disease including but not limited to symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (≥150/90mmHg) despite appropriate anti-hypertensive medication (patients with stably controlled hypertension are eligible), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvopathy requiring treatment.
* Receipt of live vaccine(s) within 30 days prior to the first dose of trial treatment.
* Other uncontrolled intercurrent illness, including but not limited to, ongoing/active infection, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events and/or compromise the ability of the patient to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemech C, Dredge K, Bampton D, Hammond E, Clouston A, Waterhouse NJ, Stanley AC, Leveque-El Mouttie L, Chojnowski GM, Haydon A, Pavlakis N, Burge M, Brown MP, Goldstein D. Phase Ib open-label, multicenter study of pixatimod, an activator of TLR9, in combination with nivolumab in subjects with microsatellite-stable metastatic colorectal cancer, metastatic pancreatic ductal adenocarcinoma and other solid tumors. J Immunother Cancer. 2023 Jan;11(1):e006136. doi: 10.1136/jitc-2022-006136. PMID 36634920

RESULTS

PARTICIPANT FLOW:
Groups:
- Pixatimod (PG545) + Nivolumab - Cohort 1: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 (MSS MCRC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
- Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 and Cohort 3: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
Period: Overall Study
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 and Cohort 3
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pixatimod (PG545) + Nivolumab: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 (MSS CRC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
- Pixatimod (PG545) + Nivolumab + Cyclophosphamide: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
- Total: Total of all reporting groups
Arm/Group | Pixatimod (PG545) + Nivolumab | Pixatimod (PG545) + Nivolumab + Cyclophosphamide | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (13.45) | 71.75 (8.26) | 66.46 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response (rate) will be expressed as the percentage of patients with Complete Response (CR) + Partial Response (PR). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD;Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Stable Disease is neither >30% shrinkage nor >20% growth of tumor.
Time Frame: Up to 26 months
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of patients
Groups:
- Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients
  Stable Disease (SD) | 40 | 37.5
  Progressive Disease (PD) | 60 | 62.5
Statistical Analysis 1: Comparison: Pixatimod (PG545) + Nivolumab - Cohort 1 vs Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3; Test type: Superiority; p = 1.0000, Fisher Exact

2. Secondary Outcome: Response Per Immune-related Response Criteria
Description: irCR (Complete Response):Disappearance of non-nodal lesions. All pathologic lymph nodes <10 mm (2 consecutive measures ≥4 weeks apart); irPR (Partial Response):≥30% decrease from baseline (2 consecutive measures ≥4 weeks apart); irPD (Progressive Disease):≥20% increase from nadir and ≥5mm (2 consecutive measures ≥4 weeks apart); irSD (Stable Disease): Not sufficient decrease for PR, nor sufficient increase for PD; irPR (Progressive Disease): Disappearance of all non-nodal lesions.All pathologic lymph nodes <10 mm (Non-Target Lesions:Any other than disappearance of all non-nodal lesions and reduction of pathologic lymph nodes <10 mm). Baseline tumor burden: sum of single diameters (short axis for nodal lesions, longest diameter for other lesions) for target lesions. In subsequent scans, the diameters of new measurable lesions are added to the tumor burden. Re-treatment: ≤5 target lesions (=/≠ original lesions) are selected and a new baseline tumor burden will be established.
Time Frame: Up to 26 months
Population: Treated patients who were radiologically evaluable for iRECIST.
Measure: Number; unit: percentage of patients
Groups:
- Pixatimod (PG545) + Nivolumab - Cohort 1: Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 (MSS CRC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients
  Unknown | 0 | 12.5
  iStable Disease | 40.0 | 37.5
  iUProgressive Disease | 60.0 | 50.0
Statistical Analysis 1: Comparison: Pixatimod (PG545) + Nivolumab - Cohort 1 vs Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3; Test type: Superiority; p = 1.0000, Fisher Exact

3. Secondary Outcome: Response Per Immune-related Response Criteria - Combined Study Population
Description: as for outcome 2
Time Frame: Up to 26 months
Population: Treated patients who were radiologically evaluable for iRECIST.
Measure: Number; unit: percentage of patients
Groups:
- Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2 & 3): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 (MSS CRC)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2 & 3)
Number analyzed (Participants) | 13
percentage of patients
  Unknown | 8
  iStable Disease | 38
  iUProgressive Disease | 54

4. Secondary Outcome: Treatment-related Adverse Events
Description: Distinct number of patients with (all-grade) related adverse events (AE), serious adverse events (SAE) and dose-limiting toxicities (DLT) if any in each cohort. Toxicity events were evaluated by NCI Common Terminology for Adverse Events (CTCAE v5.0).
Time Frame: Up to 26 months
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
participants
  Anemia | 1 | 0
  Lymphocyte count decreased | 2 | 0
  Neutrophil count decreased | 1 | 0
  Alanine aminotransferase increased | 0 | 1
  Alkaline phosphatase increased | 0 | 1
  Anorexia | 0 | 1
  Arthralgia | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Amylase increased | 0 | 1
  Fatigue | 0 | 2
  Hyperglycemia | 0 | 1
  Rash maculo-papular | 0 | 1
  Weight loss | 0 | 1

5. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of patients who remain progression-free from the initial date of treatment until 6 months afterwards, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 6 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 20 [1 to 58] | 13 [1 to 42]

6. Secondary Outcome: 1-year Progression-free Survival (PFS)
Description: Percentage of patients who remain progression-free from the initial date of treatment until 1 year afterwards, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 12 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events. | 13 [1 to 42]

7. Secondary Outcome: 2-year Progression-free Survival (PFS)
Description: Percentage of patients who remain progression-free from the initial date of treatment until 2 years afterwards, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 24 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events. | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events.

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is the time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression), whichever occurs first, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 27 months
Population: Treated patients who were radiologically evaluable.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pixatimod (PG545) + Nivolumab (Cohorts 1): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  Cohort 1 - Pixatimod (PG545) + Nivolumab - melanoma & NSCLC
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
- Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
Arm/Group | Pixatimod (PG545) + Nivolumab (Cohorts 1) | Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2)
Number analyzed (Participants) | 5 | 8
months | 2.00 [1.00 to NA] — Upper bound of CI not reached due to low number of events. | 2.00 [1.00 to NA] — Upper bound of CI not reached due to low number of events.

9. Secondary Outcome: Progression-free Survival (PFS) - Combined Study Population
Description: Percentage of patients with Progression-free survival (measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression)), whichever occurs first, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 6 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3): Pixatimod : 25 mg IV, weekly
  Nivolumab: 480 mg IV, Q4 weeks
  cyclophosphamide: 50 mg PO twice daily (Day 1-Day 7; Day 15-Day 21) with a 7-day drug free interval (Day 8-Day 14 and Day 22-Day 28)
  Cohort 1 - Pixatimod (PG545) + Nivolumab - melanoma & NSCLC and Cohort 2 (PD-1 R/R melanoma) and Cohort 3 (PD-1 R/R NSCLC)
  Pixatimod: Pixatimod is an investigational drug that is being evaluated in studies involving melanoma, non-small cell lung cancer, and microsatellite stable colorectal cancer.
  Nivolumab: Nivolumab is approved by the FDA for the treatment of melanoma, non-small cell lung cancer (NSCLC), malignant pleural mesothelioma, renal cell carcinoma, classical Hodgkin lymphoma, squamous cell carcinoma of head/neck, urothelial carcinoma, MSI-H colorectal cancer, hepatocellular carcinoma, gastric carcinoma and gastroesophageal junction (GEJ) cancer
  Cyclophosphamide (low dose): Cyclophosphamide is approved by the FDA for the treatment of acute lymphoblastic leukemia, acute monocytic leukemia, acute myeloid leukemia, breast cancer, chronic granulocytic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin lymphoma, multiple myeloma, mycosis fungoides, neuroblastoma, non-Hodgkin lymphoma, ovarian cancer, retinoblastoma. Low-dose (immunomodulatory) cyclophosphamide is being studied in combination with various types of immunotherapy including nivolumab and pembrolizumab
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 15 [2 to 39]

10. Secondary Outcome: Progression-free Survival (PFS) - Combined Study Population
Description: as for outcome 9
Time Frame: Up to 12 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 15 [2 to 39]

11. Secondary Outcome: Progression-free Survival (PFS) - Combined Study Population
Description: as for outcome 9
Time Frame: Up to 24 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events.

12. Secondary Outcome: Progression-free Survival (PFS) - Combined Study Population
Description: as for outcome 8
Time Frame: Up to 27 months
Population: Treated patients who were radiologically evaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
months | 2.00 [1.00 to 4.00]

13. Secondary Outcome: 6-month Overall Survival (OS)
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at one year.
Time Frame: Up to 6 months
Population: All trial participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 75 [13 to 96] | 50 [15 to 77]

14. Secondary Outcome: 1-year Overall Survival (OS)
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at one year.
Time Frame: Up to 12 months
Population: All trial participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events. | 19 [1 to 54]

15. Secondary Outcome: 2-year Overall Survival (OS)
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at two years.
Time Frame: Up to 24 months
Population: All trial participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 5 | 8
percentage of patients | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events. | 0 [NA to NA] — Upper and lower bound of CI not reached due to low number of events.

16. Secondary Outcome: Overall Survival (OS) - Combined Study Population
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at 6 months.
Time Frame: Up to 6 months
Population: All trial patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 61 [29 to 81]

17. Secondary Outcome: Overall Survival (OS) - Combined Study Population
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at 12 months.
Time Frame: Up to 12 months
Population: All trial patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 13 [1 to 43]

18. Secondary Outcome: Overall Survival (OS) - Combined Study Population
Description: Percentage of patients that remain alive from the start of treatment until death from any cause at 24 months.
Time Frame: Up to 24 months
Population: All trial patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
percentage of patients | 0 [NA to NA] — Not reached due to low number of events.

19. Secondary Outcome: Overall Survival (OS) - Combined Study Population
Description: The median length of time (estimated) from the start of treatment that patients remain alive, until death from any cause.
Time Frame: Up to 27 months
Population: All trial patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2, 3)
Number analyzed (Participants) | 13
months | 11.00 [4.00 to 12.00]

20. Secondary Outcome: Change in CD8+ T-cells
Description: Percent change in cellular frequency from baseline in the CD8+ T cell infiltrate and/or NK cell in the tumor and TME in tumor biopsies at treatment timepoints.
Time Frame: At baseline, 4 weeks
Population: Data not collected.
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Objective Response Rate (ORR) - Combined Study Population
Description: as for outcome 1
Time Frame: Up to 26 months
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Pixatimod (PG545) + Nivolumab or Pixatimod (PG545) + Nivolumab + Cyclophosphamide (Cohorts 1, 2 & 3)
Number analyzed (Participants) | 13
percentage of patients
  Stable Disease (SD) | 38
  Progressive Disease (PD) | 62

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events occurring up to 26 months from the date start of treatment.
Arm/Group | Pixatimod (PG545) + Nivolumab - Cohort 1 | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3
All-Cause Mortality (participants affected / at risk) | 3/5 | 6/8
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/8
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pixatimod (PG545) + Nivolumab - Cohort 1 (N=5) | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3 (N=8)
Sinus tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pixatimod (PG545) + Nivolumab - Cohort 1 (N=5) | Pixatimod (PG545) + Nivolumab + Cyclophosphamide - Cohort 2 & Cohort 3 (N=8)
Anemia (Blood and lymphatic system disorders) | 2 | 5
Blood and lymphatic system disorders - Other, specifyAmylase increased (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Cardiac disorders - Other, specifySinus Tachycardia, Intermittent (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Blurred vision (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
General disorders and administration site conditions - Other, specifyHot Flashes (General disorders) | 0 | 1
Pain (General disorders) | 1 | 3
Herpes simplex reactivation (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyInfection- other- fever, elevated lactate, joint aches (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4
Activated partial thromboplastin time prolonged (Investigations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 2
Cholesterol high (Investigations) | 1 | 1
Creatinine increased (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Weight loss (Investigations) | 0 | 3
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyKnee Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Nervous system disorders - Other, specifyNeuropathy-intermittent (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Glucosuria (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1
Renal and urinary disorders - Other, specifyUrinary Odor (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyCOVID-19 Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Vascular disorders - Other, specifyHeadache (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT05061017/Prot_SAP_000.pdf